CLINICAL TRIAL: NCT02266082
Title: Biobehavioral Predictors of Persistent Post-Surgical Pain in Women Undergoing Breast Cancer Treatment
Brief Title: Persistent Post-Surgical Pain in Women With BrCA
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400616; OCR15052 (Other: University of Florida)
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Chronic Pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A stool sample for microbiota analysis will be collected by participants at home using a standard test kit, and returned via mail. Fecal microbial DNA will be extracted from between 50-200 mg of fecal material. The 16S ribosomal gene (V4 region) of each sample will be amplified using a barcoding system to allow multiplexing with the Illumina MiSeq system.
  Blood samples will be collected to measure C-reactive protein (CRP) (at each visit) and telomerase/telomere and 25(OH)D level at baseline and the 6-month visit. Venous blood samples will be collected by trained staff.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — There is no intervention in this study.

SUMMARY:
Women with early-stage breast cancer (BrCA) are surviving longer, but many experience symptoms after curative treatments. Approximately 50% of BrCA survivors experience persistent pain post-surgery. Identifying individuals at high risk for long-term symptoms is important for restoring function and enhancing quality of life. This pilot study will investigate psychological (depression, anxiety, catastrophizing) and biological (inflammatory markers, gut microbiome, pain sensitivity) correlates of persistent post-surgical pain in women participants with early-stage BrCA. The investigators will also investigate the type of surgery that participants had and whether it is related to persistent pain. The investigators plan explore these factors over time.

DETAILED DESCRIPTION:
Subjects participate in a brief telephone or in-person screening to determine eligibility for this study. The first in-person visit to the UF Pain Clinical Research Unit (CRC) is scheduled to coincide with a pre-operative testing or a clinic visit. During this first visit, more health information is collected related to the eligibility criteria for the study and if the visit should proceed. The in-person screening process takes about 30 minutes. The Informed Consent will be reviewed to make sure that the subjects understand everything that is involved with the study. After consent, participants are randomly assigned, like the flip of a coin, a participant ID number known only to the investigators. The participants may choose not to continue or be excluded from the study after providing the screening information. The demographic and health information provided will be shredded. These names will be kept in a locked file, however, so that the investigators don't contact them again for screening. It will be indicated, next to the name and ID number, the reason for exclusion from the study. A copy of the signed informed consent form will remain in a locked file as well for documentation purposes.

If selected for this study and agree to participate, participants will be asked to complete several tests. These tests will take around 2 hours, and will be done following the screening questions during the first visit. The first visit will take about 2 ½ hours. There will be a second and third visit (approximately 3 and 6 months later) to the UF Pain CRC for follow-up testing. Each visit will last about 2 hours. Every effort will be made to combine these visits with regular post-surgery follow-up visits to the clinic or your health care provider. Each participant's hospital medical record associated with their surgery for breast cancer will be assessed for the amount of pain they experienced following their surgery and the pain medications that they received. Information related to the type of surgery (i.e., lumpectomy, mastectomy, or reconstruction), the results of the biopsies and lymph node tests, the characteristics of the breast tumor, and information about your surgery (e.g., type of anesthesia, duration of surgery, surgical complications) will be collected.

The following will occur during all 3 visits to the center. Information about health and medications will be collected. At the 2nd and 3rd visits, any changes to health and medications since the last visit will be collected. Blood pressure, heart rate, height and weight information will be collected from all participants. Surveys about participant's thoughts and feelings about pain will be conducted.

A trained professional will draw blood (about 1-2 teaspoons) from a vein your arm. This will be used to measure laboratory values associated with inflammation in the body. Specifically, the investigators will look for biomarkers, such as chemicals and hormones that might be related to pain. They will also check the level of vitamin D in your blood. No fasting is required before these blood tests. The stored blood sample will not be labeled with the participant's name. It will be labeled only with the ID number. The samples will be stored in the University of Florida Clinical and Translational Science Biorepository.

The Investigators will instruct participants in how to use a stool specimen kit. It will be used at home and returned in the mail. A stamped envelope will be provided to the participants with each kit. This will be used to measure microbes in your gut that are associated with inflammation. The stored stool sample will not be labeled with the participant's name. It will be labeled only with the ID number. The samples will be stored in a researcher's laboratory at the University of Florida. If participants are pre-menopausal woman, a urine pregnancy test may be required.

Several tests to measure sensitivity and tolerance to pain will be performed.

1. Pressure Sensation Test - applies pressure to one knee, thigh, shoulder and arm. The pressure may be slowly increased, and participants will be asked to tell the examiner when they begin to feel discomfort or mild pain. As soon as pain is felt, the pressure will be removed.
2. Mechanical Sensation Test - a handheld probe that has a small nylon tip to tap the knee and hand. The investigator will ask participants to tell how painful this feels.
3. Heat Pain Test - Sensitivity to heat pain will be tested using a commercially available sensory testing machine that is widely used in clinical settings. The machine has a small square piece that is used to apply heat to the skin. Heat will be applied to one knee and arm. The amount of heat is controlled by a computer. The procedure can be stopped at any time so that participants do not experience pain that is unacceptable.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with breast cancer (based on biopsy)
* scheduled for surgery (either lumpectomy or mastectomy, with anticipated sentinel node dissection and possible axillary lymph node dissection)
* between 40 - 75 years of age.

Exclusion Criteria:

* history of previous cancer, chemotherapy or radiation, cardiovascular or neurological conditions, bowel surgery, or hospitalization for mental illness in past year
* chronic pain conditions or daily use of opioids
* pregnant or nursing
* diagnosed with metastatic breast cancer after surgery and cancer staging is completed (post-lymph node dissection)
* any other condition that in the opinion of the principal investigator may compromise participation in this study

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with early stage breast cancer, who plan to have breast surgery at UF Health/Shands Hospital in Gainesville, Florida
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity from baseline to 3 and 6 months post-surgery | Baseline, 3 months and 6 months post-operative
  Self-reported pain intensity will be assessed using the NIH PROMIS-43 subscale for pain measurement. Pain intensity is rated on a 10 point scale, with 0 indicating no pain and 10 indicating worst pain imaginable.

SECONDARY OUTCOMES:
Persistent Pain Intensity | 1 year post-operative
  Self-reported pain intensity will be assessed using the NIH PROMIS-43 subscale for pain measurement. Pain intensity is rated on a 10 point scale, with 0 indicating no pain and 10 indicating worst pain imaginable.
Change from baseline in C-reactive protein | Baseline, 3 months and 6 months post-operative
  For the measurement of serum CRP levels, a commercially available immuno-turbidimetric assay will be used. Higher levels of CRP are associated with higher levels of systemic inflammation.
Change from baseline in Gut microbiome | Baseline, 3 months and 6 months post-operative
  The number and type of species found in the intestinal microbiota will be assessed.
Change from baseline in Vitamin D (25(OH)D) | Baseline and 6 months post-operative
  Blood samples will be collected to measure total 25(OH)D level. The results are expressed in nanograms per mililiter (ng/ml), with optimal levels ranging from 30-80 ng/ml, insufficient levels ranging from 10-29 ng/ml, and severe deficiency as less than 10 ng/ml.
Change from baseline in Telomerase | Baseline and 6 months post-operative
  Blood samples will be collected to measure telomerase. Telomerase activity is measured by evaluating the amount of inorganic pyrophosphate generated in Polymerase Chain Reaction (PCR) amplification of telomerase elongation product, with use of the sensitive enzymatic luminometric inorganic pyrophosphate detection assay (ELIDA). TRAP connected with ELIDA (TRAP-ELIDA) can quantitatively detect telomerase activity within linearity from 2 to 1000 cell equivalents.
Change from baseline in Pain Interference | Baseline, 3 months and 6 months post-operative
  Self-reported pain interference will be assessed using the NIH PROMIS-43 subscale, consisting of 6 questions. Pain interference is rated on a 5 point scale, with 1 indicating that pain does not interfere at all and 5 indicating that pain interferes with activities very much. Total scores for this subscale range from 6 to 30 (most interference).
Change from baseline in Pain Catastrophizing | Baseline, 3 months and 6 months post-operative
  The Pain Catastrophizing Scale will be used to measure pain cognitions. This 13 item scale is scored on a 0-5 scale, in which 0 indicates the thought does not occur and 5 indicates that the cognition occurs all the time. Total score ranges from 0-65.
Change from baseline in Depression | Baseline, 3 months and 6 months post-operative
  Self-reported depression will be assessed using the NIH PROMIS-43 subscale, consisting of 6 questions about depression. Responses are rated on a 5 point scale, with 1 indicating the response never occurs and 5 indicating the response always occurs. Total scores for this subscale range from 6 to 30.
Change from baseline in Anxiety | Baseline, 3 months and 6 months post-operative
  Self-reported anxiety will be assessed using the NIH PROMIS-43 subscale, consisting of 6 questions about feelings of anxiety. Responses are rated on a 5 point scale, with 1 indicating the response never occurs and 5 indicating the response always occurs. Total scores for this subscale range from 6 to 30.
Change from baseline in Pain Qualities | Baseline, 3 months and 6 months post-operative
  Characteristics of neuropathic and nociceptive pain are assessed with the Pain Qualities Scale. This consists of 20 items that rate different pain characteristics on a 0-10 scale, with 0 indicating none of that characteristic and 10 indicating the most of that characteristic.
Surgical Variables | First 48 hours post-operative
  Data about the surgical procedure will be collected from the surgical and anesthesia reports in the medical record. This will include information about surgical type (e.g., lumpectomy, mastectomy (single or double), and reconstruction. The extent of lymph node dissection (sentinel node only vs. more extensive exploration) will be recorded. The duration of surgery, type of anesthesia, amount of blood loss, and any surgical complications will also be recorded.
Change from baseline in Fatigue | Baseline, 3 months and 6 months post-operative
  Self-reported fatigue will be assessed using the NIH PROMIS-43 subscale, consisting of 6 questions about feelings of fatigue. Responses are rated on a 5 point scale, with 1 indicating the feeling occurred not at all and 5 indicating the feeling occurred very much. Total scores for this subscale range from 6 to 30.
Change from baseline in Sleep Disturbance | Baseline, 3 months and 6 months post-operative
  Self-reported sleep disturbance will be assessed using the NIH PROMIS-43 subscale, consisting of 6 questions about sleep. Overall sleep quality is rated from 1 (very poor) to 5 (very good). Responses to the remaining 5 sleep questions are rated on a 5 point scale, with 1 indicating the sleep descriptor occurred not at all and 5 indicating the sleep descriptor occurred very much. Total scores for this subscale range from 6 to 30.
Change from baseline in Physical Function | Baseline, 3 months and 6 months post-operative
  Self-reported physical disability will be assessed using the NIH PROMIS-43 subscale consisting of 6 questions. Four questions assess ability to perform daily activities, with responses scored from 1 (without any difficulty) to 5 (unable to do). Two additional question evaluate the extent to which health limits activities, with responses from 1 (not at all) to 5 (cannot do).Total scores for this subscale range from 6 to 30.
Change from baseline in Social Role Function | Baseline, 3 months and 6 months post-operative
  Self-reported ability to engage in social roles will be assessed using the NIH PROMIS-43 subscale consisting of 6 questions. Responses are scored from 1 (never has trouble/limitations) to 5 (always has trouble/limitations). Total scores for this subscale range from 6 to 30.
Acute Post-operative Pain Intensity | First 48 hours post-operative
  Self-reported acute pain intensity is rated on a 10 point Numerical rating scale, with 0 indicating no pain and 10 indicating worst pain imaginable.
Pain Treatment | First 48 hours post-operative
  All analgesic medications taken by participants preoperatively, during the first 48 hours post-operatively will be recorded.
Change from baseline in Pain Threshold and Tolerance | Baseline, 3 months and 6 months post-operative
  Quantitative Sensory Testing (QST) will be conducted to measure heat pain (warmth, threshold, tolerance), pressure pain threshold, and punctate mechanical pain (suprathreshold ratings, temporal summation). After each test, participants will rate their pain on a 0-10 scale (0 = no pain; 10 = worst pain imaginable). Scores across multiple trials of each test will be averaged to obtain a mean score.

CONTACTS AND LOCATIONS:
Overall Officials: Ann L. Horgas, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States